CLINICAL TRIAL: NCT05075811
Title: A Phase IB/IIA Study of Ossium Vertebral Bone Marrow Derived Mesenchymal Stem Cells (vBM-MSC) for the Treatment of Ileal Anal Anastomosis and Ileal Pouch Fistulas in the Setting of Crohn's Disease of the Pouch
Brief Title: Study of Ossium Mesenchymal Stem Cells for the Treatment of Pouch Fistulas in the Setting of Crohn's Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amy Lightner (Other)
Collaborators: Ossium Health, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Amy Lightner, Sponsor-Investigator, MD, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 21-860
Record Dates: First submitted 2021-09-28; First posted 2021-10-13 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Pouch, Ileal; Fistula
MeSH Terms: conditions — Fistula

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vertebral Bone Marrow Derived Mesenchymal Stem Cells (vBM-MSC) (Experimental): Direct injection of vertebral bone marrow derived mesenchymal stem cells at a dose of 100 million cells into the ileal pouch fistula(s) at baseline with a possible repeat injection at 3 months if not completely healed from the first injection.
  Interventions: Drug: Ossium vBM-MSC
- Placebo (Placebo Comparator): Direct injection of normal saline. If not completely healed after 6 months, participants will then cross over to the treatment group to receive a direct injection of vertebral allogeneic bone marrow derived mesenchymal stem cells at a dose of 100 million cells into ileal pouch fistula(s).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Ossium vBM-MSC — Vertebral bone marrow derived mesenchymal stem cells
  Other Names: Ossium Vertebral Bone Marrow Derived Mesenchymal Stem Cells
  Arms: Vertebral Bone Marrow Derived Mesenchymal Stem Cells (vBM-MSC)
Other: Placebo — Normal Saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and feasibility of using Ossium vertebral Bone Marrow Derived Mesenchymal Stem Cells (vBM-MSC) to treat people with an ileal pouch anal anastomosis (IPAA) who develop a fistula in the setting of Crohn's disease of the pouch.

DETAILED DESCRIPTION:
Proctocolectomy with ileal pouch anal anastomosis (IPAA) remains the procedure of choice for patients with ulcerative colitis (UC). IPAA allows at risk tissue to be removed with restoration of intestinal continuity while maintaining favorable long-term functional outcomes and quality of life.1 2 While less than 30% of patients experience short-term postoperative morbidity following IPAA,3-5 up to 15% of pouches will ultimately fail due to technical or inflammatory complications, the majority of which manifest as a fistula from the pouch to the perianal or vaginal locations.1,2,6-8 Pouch failure due to a fistula tract is notoriously difficult to treat. Despite immunosuppressive medications and attempts at local repair, most patients will end up with a pouch excision and permanent ostomy. This can be a devastating outcome in some patients as it impacts body image and quality of life.1

Given the high safety profile, and relative success in treating perianal disease, we sought to use a GMP grade allogeneic bone marrow derived MSCs to establish safety and secondarily monitor for healing in patients with ileal anal anastomosis and ileal pouch fistulas. This trial will use allogeneic bone marrow derived mesenchymal stem cells (MSCs) to produce regenerative signals.

This study will enroll adult men and women who have undergone IPAA at least six months prior and now have a peri-pouch fistula related to Crohn's disease of the pouch. Subjects who are refractory to conventional medical therapy will be considered. Subjects enrolled will be those that meet current indications.

ELIGIBILITY:
Inclusion Criteria

1. Men and women 18-75 years of age who have undergone an ileal pouch anal anastomosis at least 6 months prior who have developed a clinical diagnosis of Crohn's disease of the pouch as determined by a combination of clinical symptoms, pouchoscopy with biopsy, enterography.
2. Single and multi-tract (up to 2 internal and 3 external openings) fistula tract arising from the ileal pouch, ileal anal anastomosis, or anal canal distal to anastomosis that travels to the perianal skin, perineal body, or vagina. Subjects with fistulas that arise from the pouch, anastomosis, or anal canal distal to the anastomosis will both be included in enrollment. a. Acceptable internal openings and tract locations for the fistula to arise from include the ileal pouch body, the pouch anal anastomosis, and the anal canal distal to the anastomosis.

   b. Acceptable external openings and tract locations for the fistula to arise from include the perianal skin, perineal body, and/or the vaginal wall.
3. Concurrent Crohn's related therapies with stable doses (>3 months) corticosteroids, 5-ASA drugs, immunomodulators, anti-TNF therapy, anti-integrin and anti-interleukin are permitted.
4. Failed oral antibiotic therapy -any oral antibiotic that has been attempted and has not been effective for fistula closure.
5. Have failed conventional medical therapies described above, defined as a lack of response to systemic immune suppression (e.g. azathioprine, methotrexate, 6-mercaptopurine) or biologic (e.g. anti-TNF, anti-integrin, anti-interleukin) therapies to treat fistulizing CD for at least 3 months
6. Competent and able to provide written informed consent
7. Ability to comply with protocol.

Exclusion Criteria

1. Change in medical management for CD in the previous 2 months or changes anticipated in the next 2 months
2. Daily use of prednisone of greater than 20 mg per day
3. Clinically significant medical conditions within the six months before administration of vBM-MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the subject.
4. Specific exclusions;

   * HIV
   * Hepatitis B or C
5. History of cancer including melanoma (with the exception of localized skin cancers) within 1 year prior to treatment
6. Investigational drug within thirty (30) days of baseline
7. Pregnant or breast feeding or trying to become pregnant
8. Contraindications to MR evaluations: e.g. pacemaker or magnetically active metal fragments, claustrophobia
9. Unwilling to agree to use acceptable contraception methods during participation in study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Treatment related adverse events | Month 6
  Number of participants with treatment related adverse events post-injection of 100 million vertebral bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease as assessed by protocol
Complete clinical healing | Month 6
  Number of participants with complete clinical healing post-injection of 100 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease of the pouch.
  Complete Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 3 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical Healing: 100% cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Complete clinical healing | Month 12
  Number of participants with complete clinical healing post-injection of 100 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease of the pouch.
  Complete Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 3 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical Healing: 100% cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Partial healing | Month 6
  Number of participants with partial clinical healing,post-injection of 100 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Partial Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical healing: Greater than or equal to 50 % cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Partial healing | Month 12
  Number of participants with partial clinical healing,post-injection of 100 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Partial Healing is defined as:
  Radiographic Healing: MRI with an absence of a fluid collection >2 cm in 2 of 3 dimensions, lack of edema, inflammation or sign of active inflammatory response. A remnant scar of a fistula tract may remain
  Clinical healing: Greater than or equal to 50 % cessation of drainage on both clinical exam with deep palpation and per patient report and epithelization of the external fistula opening
Lack of response | Month 6
  Number of participants with lack of response post-injection of 100 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Lack of Response is defined as: Radiographic and Clinical healing which does not meet the threshold for Partial Healing
Lack of response | Month 12
  Number of participants with lack of response post-injection of 100 million allogeneic bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Lack of Response is defined as: Radiographic and Clinical healing which does not meet the threshold for Partial Healing
Worsening disease | Month 6
  Number of participants with worsening disease-injection of 100 million vertebral bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Worsening Disease is defined as:
  Radiographic: MRI with a fluid collection >2 cm in 2 of 3 dimensions, edema, inflammation or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract,
  Clinical: Increased drainage per patient report and on clinical exam
Worsening disease | Month 12
  Number of participants with worsening disease-injection of 100 million vertebral bone marrow derived MSC's for the treatment of medically refractory pouch fistulizing disease in the setting of Crohn's disease
  Worsening Disease is defined as:
  Radiographic: MRI with a fluid collection >2 cm in 2 of 3 dimensions, edema, inflammation or sign of active inflammatory response. An increased number of tracts may be seen, or increased branching from the primary tract,
  Clinical: Increased drainage per patient report and on clinical exam

CONTACTS AND LOCATIONS:
Overall Officials: Amy Lightner, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fazio VW, Kiran RP, Remzi FH, Coffey JC, Heneghan HM, Kirat HT, Manilich E, Shen B, Martin ST. Ileal pouch anal anastomosis: analysis of outcome and quality of life in 3707 patients. Ann Surg. 2013 Apr;257(4):679-85. doi: 10.1097/SLA.0b013e31827d99a2. PMID 23299522
- [Background] Ozdemir Y, Kiran RP, Erem HH, Aytac E, Gorgun E, Magnuson D, Remzi FH. Functional outcomes and complications after restorative proctocolectomy and ileal pouch anal anastomosis in the pediatric population. J Am Coll Surg. 2014 Mar;218(3):328-35. doi: 10.1016/j.jamcollsurg.2013.11.019. Epub 2013 Nov 26. PMID 24468224
- [Background] Remzi FH, Fazio VW, Kirat HT, Wu JS, Lavery IC, Kiran RP. Repeat pouch surgery by the abdominal approach safely salvages failed ileal pelvic pouch. Dis Colon Rectum. 2009 Feb;52(2):198-204. doi: 10.1007/DCR.0b013e31819ad4b6. PMID 19279412
- [Background] Foley EF, Schoetz DJ Jr, Roberts PL, Marcello PW, Murray JJ, Coller JA, Veidenheimer MC. Rediversion after ileal pouch-anal anastomosis. Causes of failures and predictors of subsequent pouch salvage. Dis Colon Rectum. 1995 Aug;38(8):793-8. doi: 10.1007/BF02049833. PMID 7634973
- [Background] Meagher AP, Farouk R, Dozois RR, Kelly KA, Pemberton JH. J ileal pouch-anal anastomosis for chronic ulcerative colitis: complications and long-term outcome in 1310 patients. Br J Surg. 1998 Jun;85(6):800-3. doi: 10.1046/j.1365-2168.1998.00689.x. PMID 9667712
- [Background] Farouk R, Pemberton JH, Wolff BG, Dozois RR, Browning S, Larson D. Functional outcomes after ileal pouch-anal anastomosis for chronic ulcerative colitis. Ann Surg. 2000 Jun;231(6):919-26. doi: 10.1097/00000658-200006000-00017. PMID 10816636